CLINICAL TRIAL: NCT06312085
Title: A Prospective, Single-arm, Non-randomized Controlled Trial to Test the Effectiveness, Safety and Performance of a Novel Dental Obturation Material
Brief Title: A Study to Assess the Clinical Success of Root Canal Treatment Using Novel Obturation Material.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lumendo AG (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EF_5301_V1.0_CIP
Record Dates: First submitted 2024-03-04; First posted 2024-03-15 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Endodontic Treatment
Keywords: Root Canal Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Endofill arm (Experimental): Endofill arm- This arm will receive the novel obturation material after root canal preparation and success of root canal treatment will be measured after 12 months
  Interventions: Device: Endofill

INTERVENTIONS:
Device: Endofill — Endofill is intended for the permanent obturation of root canals following root canal preparation and disinfection.
  Other Names: Odnefill

SUMMARY:
The goal of this study is prospective, single-arm, non-randomized controlled trial to test the effectiveness, safety and performance of a novel dental obturation material. The main question sit answers is

1. To test the effectiveness of the Endofill device for root canal obturation up to 12-month follow-up period.
2. To test the performance of the Endofill device evaluated with periapical radiographs immediately on completion of procedure.

The participants requiring root canal treatment will be treated with obturated using Endofill material and post-treatment follow-up vistis will be conducted for 1 year. This is a single-arm study with no comparison groups.

DETAILED DESCRIPTION:
Study Title:

"A prospective, single-arm, non-randomized controlled trial to test the effectiveness, safety and performance of a novel dental obturation material."

Protocol Version and Date: Version 1.0 25 May 2023

Device Risk Category: Risk category: Class IIa, Rule 8 - medium risk device (according to EU MDR).

Background and Rationale:

Endofill (EF) is a low-viscosity, injectable, hydrophilic, light- curable endodontic sealer. It is an easy-to-use, single- material root canal obturation solution that circumvents the disadvantages of existing products, thus improving ease of handling and treatment time while maintaining the clinical outcome of root canal treatments at the level of state-of-the- art treatment methods.

Endofill is used after a conventional access cavity preparation, glide path preparation, determination of the working length, cleaning/shaping of a root canal with a suitable device and irrigating/disinfecting the canal with an irrigant solution.

Endofill has undergone pre-clinical testing and is a safe product. The benefits and risks of this investigational device shall be elaborated in the protocol.

Primary objectives:

To test the effectiveness of the Endofill device for root canal obturation up to 12-month follow-up period.

To test the performance of the Endofill device evaluated with periapical radiographs immediately on completion of procedure.

Secondary objectives:

To test the safety and effectiveness, of the Endofill device by evaluating the incidence of re-treatment cases up to a 12-month follow-up period.

Primary endpoints Primary effectiveness endpoint: To measure overall healing, through rate of reduction in apical periodontitis, from baseline up to 12 months post-procedure by measuring periapical radiolucency size.

Success is measured by the PAI (periapical index) scores which will be recorded at 3m, 6m and 12 months. Success is defined as either a fully healed lesion (i.e., with no periapical radiolucency visible on the radiograph at 12 month follow up) or a healing lesion (i.e., the periapical radiolucency has decreased in size at 12 month follow up compared to pre-procedure radiographic lesion size); with no clinical symptoms such as pain or swelling.

Performance endpoint:

To measure the successful and complete obturation of root canal measured by examining the periapical radiograph taken immediately after obturation.

Secondary endpoints:

Safety endpoint: To measure freedom from postoperative pain from completion of procedure up to 1 months of follow-up (FU) period (24 hours, 48 hours, 72 hours, 7 days, and 1 month). Pain is measured by VAS assessment.

Secondary effectiveness endpoint:

Successful healing of periapical lesion up to 12 months post-procedure. Long-term effectiveness success shall be defined as a continued reduction or complete absence of periapical lesion radiolucency at 12m follow up since procedure with no clinical symptoms (i.e no discomfort in treated tooth and no percussive pain during examination)

Device failure shall be defined as root canal re-treatment or extraction requirement due to the treatment itself as the cause of failure, up to 12m post procedure along with persistence of clinical symptoms.

The study involves a safety check at 3 months' time point post-procedure. This check will be performed on the first 10 subjects to assess the safety, effectiveness, and performance of the evaluated device.

A total of 63 subjects aged 18 years and above shall be included in this study. Study Procedure

* Subjects will be selected based on inclusion and exclusion criteria and subjects will be assigned a subject ID code for the study.
* Each subject shall receive the endodontic treatment as laid out in this protocol.
* Subject dropout is addressed in the statistical analysis plan.
* The follow-up period (up to 12 months) shall permit the demonstration of clinical effectiveness, performance and safety over a period of time sufficient to represent a realistic test of the investigational device and allow any risks associated with adverse device effects to be identified and assessed.

The planned enrollment period is 6-9 months. The total expected duration of the clinical investigation is 2 - 2.5 years.

Statistical Considerations:

Full details of the analyses will be discussed in a separate statistical analysis plan (SAP). Briefly, the following endpoints will be analyzed:

Primary endpoints are

* A reduction in PAI at 12 months compared to baseline. The rate seen will be compared to a target rate of 0.85 using a non-inferiority test at a margin of 0.2.
* Successful obturation of the root canal at procedure's completion. The rate will be reported with its 95% Clopper-Pearson CI.

The secondary endpoints are

* Experiencing different levels of postoperative pain (none, mild, moderate, and severe) at 24 hours, 48 hours, 72 hours, 7 days, 1 month after the procedure. The rates will be reported with their 95% Clopper-Pearson confidence intervals.
* Root canal re-treatment in tooth treated with Endofill at 12 months post-procedure. The rate will be reported with its 95% Clopper-Pearson confidence interval.
* Duration of the obturation procedure. Summary statistics (mean, median, max, min, IQR, and range) will be reported.

Questionnaire about the quality and usability of the device.

· Summary statistics of results will be reported.

Sample Size In order to be able to establish non-inferiority within a margin of 0.2 of the target rates of 0.85, a two-sided, 95% confidence interval for the healing rate must lie above 0.85 - 0.2 = 0.65. Assuming a pessimistic scenario where the true underlying healing rate of the Endofill device is 0.02 lower than the target rate of 0.85 (i.e., 0.83), data from 56 participants are needed. This yields a power of 80% for the study. Assuming a 10% drop out rate at 12 months, the required sample size is 63.

ELIGIBILITY:
Inclusion Criteria:

• Patients aged 18-75 years with ASA (American Society of Anesthesiologists) classification 1 and 2.

ASA 1: A normal healthy patient. Example: Fit, non-obese BMI (Body Mass Index) under 30, a non-smoking patient with good exercise tolerance.

ASA 2: A patient with mild systemic disease. Example: Patient with no functional limitations and a well-controlled disease (e.g., treated hypertension, obesity with BMI under 35, frequent social drinker, or cigarette smoker).

* Patients who agreed to participate and who have signed the informed consent.
* Patients presenting with symptomatic and/or asymptomatic apical periodontitis and radiographic evidence of apical periodontitis in anterior or posterior teeth larger than 1.5 mm in diameter.
* Mature tooth with closed apices.
* Tooth that has never been treated with root canal therapy.

Exclusion Criteria:

* Patients who have pre-existing health or oral conditions that placed them at risk during the trial.
* Patients with generalized untreated periodontal disease.
* Patients with a history of analgesic intake within the past 3 days or antibiotics in the last 1 month.
* Uncooperative patients.
* Teeth with immature apices, root resorption, or requiring extensive prosthetic rehabilitation.
* Teeth that cannot be made functional nor restored or difficult to access teeth with no importance (wisdom teeth).
* Teeth with insufficient periodontal support.
* Teeth with poor prognosis for root canal treatment, for example due to deep root caries, large root resorption or open apex cases.
* Fractured teeth
* Local anatomical factors such as an inaccessible root end
* Presence of fractured instrument in the root canal
* Pregnant women
* Patients unable to understand the study procedure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of root canal treatment using Endofill | 12 months
  To measure effectiveness by assessing overall healing, through rate of reduction in apical periodontitis, from baseline up to 12 months post-procedure by measuring periapical radiolucency size.

SECONDARY OUTCOMES:
Safety of root canal treatment using endofill | 1 month
  To measure safety by measuring postoperative pain from completion of the procedure up to 1 month of follow-up period (24 hours, 48 hours, 72 hours, 7 days, and 1 month). Pain is measured by VAS assessment. It consists of a line, approximately 10 cm in length, with the left side signifying no pain with a smiling face image and the right side signifying the worst pain with a frowning face image. A patient is asked to indicate his/her perceived pain intensity along a 100 mm horizontal line, and this rating is then measured from the left edge. A VAS score of 0 indicates no pain and a score of 10 indicates the highest level of pain experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Tan Firat Eyuboglu, Prof. Dr., Principal Investigator — Medipol University
Locations (1):
- Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No